CLINICAL TRIAL: NCT05691062
Title: A Prospective, Randomized Comparison of Titanium vs. PEEK Fusion Devices in 1 Level TLIF
Brief Title: Titanium vs. PEEK Fusion Devices in 1 Level TLIF
Acronym: TLIF
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Twin Cities Spine Center (Other)
Responsible Party: Principal Investigator, Bayard Carlson, Staff Surgeon, Twin Cities Spine Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1944564
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Spine Fusion; Lumbar Spondylolisthesis; Lumbar Stenosis
MeSH Terms: conditions — Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial with two cohorts.
Who Masked: Participant
Masking Description: Subjects will be blinded to fusion device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PEEK (Experimental): Medtronic Capstone
  Interventions: Device: PEEK Fusion Device
- Titanium (Experimental): Medtronic Adaptix
  Interventions: Device: Titanium Fusion Device

INTERVENTIONS:
Device: Titanium Fusion Device — Titanium fusion device will be utilized for one-level lumbar fusion.
  Arms: Titanium
Device: PEEK Fusion Device — PEEK fusion device will be utilized for one-level lumbar fusion.
  Arms: PEEK

SUMMARY:
The objective of this study is to evaluate and follow the clinical and radiographic outcomes of patients undergoing 1 level TLIF randomized to either a titanium or a PEEK spacer to 24 months after surgery.

DETAILED DESCRIPTION:
Transforaminal lumbar interbody fusion (TLIF) remains a common surgical technique for the management of lumbar spondylosis requiring decompression and fusion. The choice of interbody spacer remains dependent on surgeon preference with a variety of options available for use. Two of the most commonly used interbody spacers are made of polyetheretherketone (PEEK) and titanium.1 While both spacers have produced reliable rates of fusion with good clinical outcomes, debate remains as to which interbody spacer is superior. Proponents of PEEK argue that it is radiolucent and has an elastic modulus similar to bone thus decreasing rates of subsidence. However, PEEK is a hydrophobic material that does not integrate with bone. Titanium on the other hand demonstrates osseointegration and may lead to increased rates of fusion.While there are retrospective studies available comparing the two materials, the studies are small and there is a paucity of prospective data comparing the radiographic and clinical outcomes of these spacers. Given the frequency with which these spacers are used, it is important to determine which spacer produces better clinical and radiographic outcomes for patients.

ELIGIBILITY:
Inclusion Criteria

1. Patients undergoing 1 level TLIF for the treatment of lumbar stenosis and spondylolisthesis who have failed at least 6 weeks of non-operative treatment.
2. Patients between 18-70 years of age at the time of surgery.

Exclusion Criteria

1. Patients under 18 or over 70 years of age at the time of surgery.
2. Patients undergoing more than 1 level of surgery.
3. Patients who have had prior lumbar fusion.
4. Patients requiring surgery for the management of infection, tumor, or trauma.
5. Patients who are pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Fusion Status of 1 level Lumbar TLIF | 12 months Post-Op
  Assess fusion status of 1 level Lumbar TLIF by reviewing patient CT Scan completed for study purposes.
Revision Surgeries | Up to 24 months Post-op
  Monitor and Record Complications and Revision Surgeries

SECONDARY OUTCOMES:
Patient Reported Outcome Measures | Preoperative time frame up to 24 months Post-op
  Data collected from patient self reported outcome tools

CONTACTS AND LOCATIONS:
Locations (1):
- Twin Cities Spine Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rickert M, Fleege C, Tarhan T, Schreiner S, Makowski MR, Rauschmann M, Arabmotlagh M. Transforaminal lumbar interbody fusion using polyetheretherketone oblique cages with and without a titanium coating: a randomised clinical pilot study. Bone Joint J. 2017 Oct;99-B(10):1366-1372. doi: 10.1302/0301-620X.99B10.BJJ-2016-1292.R2. PMID 28963159
- [Background] Hasegawa T, Ushirozako H, Shigeto E, Ohba T, Oba H, Mukaiyama K, Shimizu S, Yamato Y, Ide K, Shibata Y, Ojima T, Takahashi J, Haro H, Matsuyama Y. The Titanium-coated PEEK Cage Maintains Better Bone Fusion With the Endplate Than the PEEK Cage 6 Months After PLIF Surgery: A Multicenter, Prospective, Randomized Study. Spine (Phila Pa 1976). 2020 Aug 1;45(15):E892-E902. doi: 10.1097/BRS.0000000000003464. PMID 32675599
- [Background] Villavicencio AT, Nelson EL, Rajpal S, Beasley K, Burneikiene S. Prospective, randomized, double-blinded clinical trial comparing PEEK and allograft spacers in patients undergoing transforaminal lumbar interbody fusion surgeries. Spine J. 2022 Jan;22(1):84-94. doi: 10.1016/j.spinee.2021.06.005. Epub 2021 Jun 8. PMID 34116214
- [Background] Seaman S, Kerezoudis P, Bydon M, Torner JC, Hitchon PW. Titanium vs. polyetheretherketone (PEEK) interbody fusion: Meta-analysis and review of the literature. J Clin Neurosci. 2017 Oct;44:23-29. doi: 10.1016/j.jocn.2017.06.062. Epub 2017 Jul 21. PMID 28736113
- [Background] Cuzzocrea F, Ivone A, Jannelli E, Fioruzzi A, Ferranti E, Vanelli R, Benazzo F. PEEK versus metal cages in posterior lumbar interbody fusion: a clinical and radiological comparative study. Musculoskelet Surg. 2019 Dec;103(3):237-241. doi: 10.1007/s12306-018-0580-6. Epub 2018 Dec 10. PMID 30536223
- [Background] Nemoto O, Asazuma T, Yato Y, Imabayashi H, Yasuoka H, Fujikawa A. Comparison of fusion rates following transforaminal lumbar interbody fusion using polyetheretherketone cages or titanium cages with transpedicular instrumentation. Eur Spine J. 2014 Oct;23(10):2150-5. doi: 10.1007/s00586-014-3466-9. Epub 2014 Jul 12. PMID 25015180